CLINICAL TRIAL: NCT04709276
Title: A Phase II, Single Arm Study of Chemoimmunotherapy for the Treatment of Men With Neuroendocrine or Aggressive Variant Metastatic Prostate Cancer (CHAMP)
Brief Title: A Study of Chemoimmunotherapy for the Treatment of Men With Neuroendocrine or Aggressive Variant Metastatic Prostate Cancer
Acronym: CHAMP
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Andrew J. Armstrong, MD (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Andrew J. Armstrong, MD, Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00106278; CA209-63X (Other: Bristol Myers Squibb)
Record Dates: First submitted 2021-01-12; First posted 2021-01-14 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Prostate Neuroendocrine Carcinoma; Metastatic Prostate Cancer
Keywords: Neuroendocrine Prostate Cancer; Aggressive Variant Prostate Cancer; Chemoimmunotherapy; Nivolumab; Ipilimumab; Carboplatin; Cabazitaxel
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Nivolumab; Ipilimumab; CTLA-4 Antigen; Carboplatin; cabazitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neuroendocrine Prostate Cancer (NEPC) or Aggressive Variant Prostate Cancer (AVPC) (Experimental): Subjects with neuroendocrine prostate cancer (NEPC) or aggressive variant prostate cancer (AVPC) will receive a combination of nivolumab, ipilimumab, carboplatin and cabazitaxel for up to 10 cycles of 21 days each. After carboplatin and cabazitaxel are discontinued, a combination of nivolumab and ipilimumab will be administered.
  Nivolumab will be administered intravenously at a dose of 360 mg every 3 weeks.
  Ipilimumab will be administered intravenously at a dose of 1 mg/kg every 6 weeks.
  Carboplatin will be administered intravenously at a dose of AUC 4 mg/ml per minute.
  Cabazitaxel will be administered intravenously at a dose of 20 or 25 mg/m2.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab; Drug: Carboplatin; Drug: Cabazitaxel

INTERVENTIONS:
Drug: Nivolumab — 360 mg intravenously every 3 weeks
  Other Names: BMS-936558; MDX1106; ONO-4538
Drug: Ipilimumab — 1 mg/kg intravenously every 6 weeks
  Other Names: BMS-734016; MDX010; MDX-CTLA4
Drug: Carboplatin — AUC 4 mg/ml per minute intravenously every 3 weeks for up to 10 cycles.
  Subjects will also receive granulocyte-colony stimulating factor (G-CSF) therapy while receiving carboplatin.
Drug: Cabazitaxel — 20 or 25 mg/m2 intravenously every 3 weeks for up to 10 cycles.
  Subjects will also take prednisone by mouth at a dose of 10 mg daily and receive granulocyte-colony stimulating factor (G-CSF) therapy while receiving cabazitaxel.
  Other Names: JEVTANA

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of a combination of nivolumab, ipilimumab, cabazitaxel and carboplatin in men with neuroendocrine prostate cancer (NEPC) or other aggressive variants of prostate cancer (AVPC). This study will also investigate biomarkers to gain a better understanding of how the drug combination of nivolumab, ipilimumab, cabazitaxel and carboplatin affects these types of prostate cancer and the immune system. Eligible subjects will receive up to 10 cycles of nivolumab, ipilimumab, carboplatin and cabazitaxel followed by maintenance nivolumab and ipilimumab. Subjects may continue receiving study drugs until cancer progression, severe toxicity, withdrawal of consent, 3 years from the initial dose of study drugs or study termination, whichever occurs earlier. Subjects will be followed for 3 years from the initial dose of study drugs.

ELIGIBILITY:
Inclusion Criteria:

1. Neuroendocrine-like prostate cancer, based on histology OR based on clinical presentation as defined by meeting one of the two below criteria. All subjects must submit their primary tumor or metastatic biopsy pathology specimens to the Duke Cancer Institute where they will be centrally reviewed by Duke Pathology. Central Duke pathologic review is not required for screening but rather for confirmation of histologic subtype. Local pathologic review is sufficient for eligibility determination.

   1. Criterion 1: Presence of 1 of 3 histologically proven diagnoses: 1) Primary small cell carcinoma of the prostate, defined by classic histologic features such as small tumor cells with scanty cytoplasm, darkly stained nuclei with homogeneous chromatin pattern. The tumor cells do not form glandular structure but grow as solid sheets with frequent mitotic figures and necrosis; 2) Intermediate atypical carcinoma of the prostate, which has histologic features distinct from small cell carcinoma or adenocarcinoma. The tumor grows as solid sheets or vague glandular structures. The tumor cells have moderate amounts of cytoplasm and centrally located, round and regular nuclei with fine, granular and homogeneous chromatin. Mitosis and necrosis are absent; 3) mixed histology tumors of the prostate, containing both adenocarcinoma and neuroendocrine or small cell components.
   2. Criterion 2: Presence of histologically proven adenocarcinoma of the prostate without any sign of neuroendocrine or small cell histology that is radiographically progressing with the following poor risk features:

   i. Prior progression despite therapy with abiraterone acetate, darolutamide or apalutamide and/or enzalutamide.

   ii. At least one of the following: 1) Visceral metastases; 2) Low PSA (<10 ng/mL) with either A. bulky lymphadenopathy or pelvic mass (>5 cm) or B. high volume (>20) bone metastases; 3) Short interval (<6mo) to CRPC following initiation of hormonal therapy 4) Pathogenic alterations in two of three genes: TP53, RB1, and PTEN. 5) Predominantly lytic bone metastases on imaging, 6) Presence of neuroendocrine markers on histology (positive staining of chromogranin A or synaptophysin) or in serum (abnormal high serum levels for chromogranin A or gastrin releasing peptide (GRP)) at initial diagnosis or at progression; 7) Any of the following in the absence of other causes: A. elevated serum LDH (>= IULN); B. malignant hypercalcemia; C. elevated serum CEA (>2x IULN).
2. Available archival tumor tissue for pathologic review and correlative studies. Tumor tissue (localized or metastatic) does not need to be received but rather identified and available (slides and/or blocks) to be sent to Duke.
3. Documented progressive metastatic CRPC as determined by the provider based on at least one of the following criteria:

   1. PSA progression defined as 25% increase over baseline value with an increase in the absolute value of at least 2.0 ng/mL that is confirmed by another PSA level with a minimum of a 1 week interval and a minimum PSA of 2.0 ng/mL. Note: If confirmed rise is the only indication of progression, a minimal starting value of 1.0 ng/mL is acceptable, unless pure small-cell carcinoma.
   2. Soft-tissue progression based on new lesions or growth of existing soft tissue metastases.
   3. Progression of bone metastasis with one or more new bone lesion(s) by imaging.
4. Castrate levels of serum total testosterone (<50 ng/dl) OR ongoing documented ADT.

   a. These criteria are not required when pure small cell prostate cancer is present.
5. Karnofsky performance status of 70 or higher.
6. Acceptable initial laboratory values within 14 days of Cycle 1 Day 1
7. Age >18
8. Subjects with a partner who is a woman of child-bearing potential must agree to use one form of highly effective contraception as detailed in Section 8.3 of this protocol during the treatment period with cabazitaxel. Subjects receiving cabazitaxel or nivolumab must also refrain from donating sperm during this period.
9. Willing and able to provide written informed consent and HIPAA authorization for the release of personal health information.
10. Life expectancy of over 3 months as determined by treating physician.

Exclusion Criteria:

1. Has received prior therapy for prostate cancer with abiraterone or androgen receptor antagonists (e.g. enzalutamide darolutamide, apalutamide) within two weeks of study treatment initiation.
2. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137).
3. Has received other prior systemic anti-cancer therapy not otherwise addressed by other eligibility criteria including investigational agents within 4 weeks prior to study treatment initiation
4. Prior receipt of cabazitaxel chemotherapy or 2 or more chemotherapy regimens in the mCRPC setting.
5. Has received prior radiotherapy within 2 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
6. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
7. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention.
8. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
9. Has a history of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 2 years.
10. Has known active untreated CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment greater than prednisone 10mg (or equivalent) for at least 14 days prior to first dose of study intervention.
11. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
12. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
13. Has an active infection requiring systemic therapy.
14. Has a known uncontrolled Human Immunodeficiency Virus (HIV) infection based on detectable HIV viral load and abnormal CD4 count of <350/mm3.
15. Has a known active Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection.
16. Has a known active TB (Bacillus Tuberculosis) infection.
17. Has ≥ Grade 2 neuropathy.
18. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
19. Has known current psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
20. Has had an allogenic tissue/solid organ transplant.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects who are progression-free and alive (progression-free survival) at 6 months | 6 months
  Progression-free survival will be determined by immune modified or Prostate Cancer Working Group 3 (PCWG3)-defined RECIST 1.1 radiographic criteria.

SECONDARY OUTCOMES:
Proportion of subjects who are progression-free and alive (progression-free survival) at 12 months | 12 months
  Progression-free survival will be determined by immune modified or PCWG3-defined RECIST 1.1 radiographic criteria.
Proportion of subjects who are progression-free and alive (progression-free survival) and without severe toxicity leading to treatment discontinuation at 6 and 12 months | 6 and 12 months
  Progression-free survival will be determined by immune modified or PCWG3-defined RECIST 1.1 radiographic criteria.
Overall survival | 6, 12 and 24 months
Median overall survival | Through study completion (up to 3 years)
Describe the radiographic progression free survival (rPFS) | Through study completion (up to 3 years)
  Radiographic progression free survival will be determined by immune modified PCWG3-defined RECIST criteria.
Describe the best radiographic response by immune modified PCWG3-defined RECIST radiographic response. | Through study completion (up to 3 years)
  Radiographic response will be determined by immune modified PCWG3-defined RECIST criteria.
Describe the toxicities of nivolumab, and ipilimumab in combination with carboplatin and cabazitaxel using NCI CTC v5.0. | Through discontinuation of carboplatin and cabazitaxel dosing (up to 30 weeks)
  The toxicity and safety will be graded using NCI CTCAE v5.0.
Describe the changes in the blood-based biomarker Prostate-Specific Antigen (PSA) over time | Through discontinuation of study drugs (up to 3 years)
  PSA
Describe the changes in the blood-based biomarker chromogranin-A over time | Through discontinuation of study drugs (up to 3 years)
  chromogranin-A
Describe the changes in the blood-based biomarker carcinoembryonic antigen (CEA) over time | Through discontinuation of study drugs (up to 3 years)
  CEA
Describe the changes in the blood-based biomarker lactate dehydrogenase (LDH) over time | Through discontinuation of study drugs (up to 3 years)
  LDH
Describe the changes in the blood-based biomarker alkaline phosphatase over time | Through discontinuation of study drugs (up to 3 years)
  alkaline phosphatase

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Armstrong, MD, ScM, Principal Investigator — Duke University
Locations (3):
- United States (3):
  - Weill Cornell Medicine, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No